CLINICAL TRIAL: NCT03218007
Title: A 2A Receptor (A2 AR) as a Novel Biomarkers for Physician Decision-making Improvement Evaluation's Patients With Suspected Acute Coronary Syndrome But Negative Troponin.
Brief Title: A2 AR as a Novel Biomarkers for Physician Decision-making Improvement Evaluation's Patients With Suspected Acute Coronary Syndrome But Negative Troponin.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2017-36; 2017-A01836-47 (Other: idrcb)
Record Dates: First submitted 2017-06-30; First posted 2017-07-14 (Actual); Last update posted 2021-10-12 (Actual); Status verified 2020-10

CONDITIONS: Acute Coronary Syndrome
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- acute coronary syndrome (Experimental)
  Interventions: Biological: blood samples

INTERVENTIONS:
Biological: blood samples — to evaluate expression and functionnaly activity of A2AR

SUMMARY:
One proposed strategy is the stratification of troponin-negative patients with biomarker testing at presentation to facilitate the clinically-appropriate rapid discharge from the emergency department of patients who present with low-intermediate risk chest pain, and conversely to triage appropriate Non sustained ST elevation acute coronary syndrome (NSTE-ACS) patients to Cardiology beds, stress and non-invasive imaging modalities. Biomarkers such as high-sensitivity troponin (hs-cTn), heart-type fatty acid-binding protein (H-FABP), CRP, brain natriuretic peptide (BNP); and copeptin and ischemia-modified albumin are an important advance for diagnostic testing for ACS (4). Regarding novel biomarker testing at presentation, the addition of these biomarkers demonstrated increased sensitivity at an acceptable QALY threshold, but more evidence is needed (5,6). A reliable method for the diagnosis of minimal cardiac ischemia would meet a strong demand for the sensitive diagnosis of coronary artery disease in patients with chest pain but unremarkable ECGs and biomarkers. Adenosine is an endogenous nucleoside cardioprotective agent. Its cardiovascular effects are mediated throught the activation of A2A Receptor (A2 AR) and play a major role in the regulation of Coronary flow CF. As altered coronary blood flow occurs in patients with CAD, it has been showed that that A2AR expression and functional activity play a role in CAD. In a previous studies the team have developped an agonist-like monoclonal antibody to study expression level of this receptor and their functional activity. Recently , Gariboldi demonstrated that measuring the expression level of A2AR on peripheral blood mononuclear cells ( PBMC) represents a good tool to address in situ expression in coronary tissues of CAD patients.

DETAILED DESCRIPTION:
In the diagnostic setting of ACS, expression and functionnaly activity of A2AR could be a sensitive detection method for ischemia. It would be a powerful tool for risk stratification of patients presenting with chest pain but unremarkable ECG and blood tests. the investigateors therefore designed a blind multicentrique prospective study to evaluate expression and functionnaly activity of A2AR in the management of undifferentiated chest pain The objective of the study was to evaluate diagnostic accuracy between this novel biomarkers A2AR and invasive and non -invasive evaluation of patients with suspected coronary artery disease (CAD).

ELIGIBILITY:
Inclusion Criteria:

* A subject with a symptomatology consistent with acute coronary syndrome for at least 15 min and less than 6 hours (eg discomfort, tightness or chest pain, pain radiating to the left arm or both arms, pain in the jaw, Pain in the back / neck / stomach, dyspnea, cold sweats, nausea / vomiting, dizziness)
* Man or woman,
* over 18 years,
* Patient agreeing to participate in the study and having signed informed consent.

Exclusion Criteria:

* Minor Patient
* Patient not having signed informed consent (refusal, physical or mental incapacity ...) --Patient with an evolutive septic process, neoplasia undergoing treatment, dialysed renal insufficiency, history of surgery or coronary angioplasty less than six months old.

Cardiac, renal or hepatic transplantation

* elevation of troponin
* Cardiac arrest
* A subject whose symptomatology clearly eliminates acute coronary syndrome (penetrating trauma, traumatic lesion by crushing ...)
* Patient who died between the time of inclusion and arrival in cardiology intensive care (ICU)
* Patient withdrawing consent during study
* Vulnerable people unable to fully integrate the objectives, benefits and risks of research and to give their informed consent
* Pregnant women
* Persons deprived of their liberty
* Persons admitted to health and social facilities for therapeutic purposes
* Protected persons

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2017-11-10 (Actual); Primary Completion 2019-05-15 (Actual); Study Completion 2019-05-15 (Actual)

PRIMARY OUTCOMES:
dosage of adenosine | 12 MONTHS
  evaluate expression and functionnaly activity of A2AR

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Olivier ARNAUD, Study Director — Assistance Publique Hopitaux De Marseille
Locations (1):
- Assistance Publique Hopitaux de Marseille, Marseille, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Paganelli F, Resseguier N, Marlinge M, Laine M, Malergue F, Kipson N, Armangau P, Pezzoli N, Kerbaul F, Bonello L, Mottola G, Fenouillet E, Guieu R, Ruf J. Specific Pharmacological Profile of A2A Adenosine Receptor Predicts Reduced Fractional Flow Reserve in Patients With Suspected Coronary Artery Disease. J Am Heart Assoc. 2018 Apr 13;7(8):e008290. doi: 10.1161/JAHA.117.008290. PMID 29654194